CLINICAL TRIAL: NCT02512289
Title: Impact of Non-invasive Brain Stimulation, Associated With Upper Limb Robot-assisted Therapy, on Motor Recuperation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Collaborators: University Hospital of Mont-Godinne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IONS-Gilliaux-03
Record Dates: First submitted 2014-08-25; First posted 2015-07-30 (Estimated); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Real stimulation (Active Comparator): real tDCS associated with robot-assisted therapy (RAT)
  Interventions: Device: tDCS (ELDITH) and RAT (REAplan)
- Sham stimulation (Sham Comparator): Sham tDCS associated with RAT
  Interventions: Device: tDCS (ELDITH) and RAT (REAplan)

INTERVENTIONS:
Device: tDCS (ELDITH) and RAT (REAplan) — Transcranial direct-current stimulation( ELDITH) and Robot-assisted therapy by using REAplan

SUMMARY:
tDCS (transcranial direct current stimulation) and robot assisted therapy (RAT) will be used in chronic stroke patients to improve a variety of functions with upper limb.

DETAILED DESCRIPTION:
tDCS and RAT will be used in chronic stroke patients to improve a variety of functions such as motor functions with upper limb.

tDCS will be applied in a placebo-controlled, double-blind, randomised fashion. A session of RAT will be associated with tDCS/placebo. Behavioural data will be collected before and after tDCS, associated with RAT.

ELIGIBILITY:
Inclusion Criteria:

* stroke with at least slight deficit in upper limb

Exclusion Criteria:

* epilepsy
* contraindication to tDCS
* presence of metal in the head
* inability to understand/complete behavioural tasks
* chronic intake of alcohol or recreative drugs
* major health condition (e.g. terminal renal failure, instable heart failure etc …)
* pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-01-09; Primary Completion 2014-01-09 (Actual); Study Completion 2015-07-30 (Actual)

PRIMARY OUTCOMES:
Upper Limb Kinematics | kinematic assessment of the upper limb at Baseline (>6 months after stroke), immediately after intervention (20min of tDCS+RAT)

SECONDARY OUTCOMES:
Box and Block test | Manual dexterity assessment at Baseline (>6 months after stroke), immediately after intervention (20min of tDCS+RAT)
Purdue Pegboard Test | Digital dexterity assessment at Baseline (>6 months after stroke), immediately after intervention (20min of tDCS+RAT)

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Lejeune, Professor, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (2):
- Belgium (2):
  - Cliniques Universitaires Saint Luc, Brussels
  - CHU Dinant-Godinne UCL, Mont Godinne